CLINICAL TRIAL: NCT03888690
Title: Randomized Controlled Trial Evaluating the Effectiveness of the Virtual Reality Distraction Compared to Current Practice, on Reducing Procedural Pain in Children and Adolescents Supported in Pediatric Onco-Hematology Unit.
Brief Title: Effect of Virtual Reality Distraction on Procedural Pain for Children and Adolescents in Onco-Hematology Unit.
Acronym: ReVaDo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRU NANCY
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Procedural Pain; Procedural Anxiety; Virtual Reality
Keywords: Children; Adolescent; non pharmacological interventions; onco-hematologic
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Interventional monocentric regional study opened in crossover test with randomization of sequence (sequence 1 "with then without Virtual Reality", sequence 2 "without then with Virtual reality").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With and then without VR (Active Comparator): Virtual Reality with standardized procedures for first intervention, Standardized procedures for second intervention, without VR.
  Interventions: Device: Virtual Reality Headset
- Without and then with VR (Active Comparator): Standardized procedures without VR for first intervention, Virtual Reality with standardized procedures for second intervention.
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Standardized procedures, with or without Virtual Reality Headset.

SUMMARY:
* Demonstrate the effectiveness of the Virtual Reality (VR) distraction on pain reduction in children and adolescents in onco-hematology unit compared to standard practice.
* Evaluate the impact of VR on the level of anxiety induced by invasive procedures
* Report traceability of assessment of pain and anxiety scores, and reproducibility of procedural analgesia techniques.
* Evaluate the impact of VR on the short-term consequences of procedural pain, especially in terms of phobia of care.

DETAILED DESCRIPTION:
Diagnosis and therapeutic management of onco-hematological pathologies in children and adolescents require multiple invasive procedures that cause pain and discomfort. These are paramedical procedures (blood sampling on the peripheral vein, placement of infusions, placement of Hubert's needles on an implantable device, ...) and medical procedures (lumbar punctures, medullary punctures, ...).

The short-term (phobia of care) and long-term consequences (memory of pain, behavioral disorders, nociceptive sensitization) are clearly reported in the medical literature, and the importance of thinking about pharmacological and non-pharmacological techniques well-established procedural pain prevention.

The quality of the management of the pain and anxiety induced by these invasive oprocedures in pediatric onco-hematology conditions the adhesion to the care and the treatments, and thus constitutes a challenge in the care of the patients. The non-pharmacological methods are numerous and still insufficiently used by the care teams. Virtual Reality is on interesting option.

ELIGIBILITY:
Inclusion Criteria:

* Children or Adolescent supported in onco-hematologic unit.

Exclusion Criteria:

* Serious behavioral disorders
* Serious neurosensory deficit

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 1 hour
  Analogical visual scale

SECONDARY OUTCOMES:
Anxiety scores | 1 hour
  Yale scale
Traceability of the procedure | 12 months
  Pain management scorecard

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic MANSUY, Principal Investigator — CHRU NANCY
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, Lorraine, France

REFERENCES:
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Result] Felluga M, Rabach I, Minute M, Montico M, Giorgi R, Lonciari I, Taddio A, Barbi E. A quasi randomized-controlled trial to evaluate the effectiveness of clowntherapy on children's anxiety and pain levels in emergency department. Eur J Pediatr. 2016 May;175(5):645-50. doi: 10.1007/s00431-015-2688-0. Epub 2016 Jan 12. PMID 26755209
- [Result] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Result] Aydin D, Sahiner NC, Ciftci EK. Comparison of the effectiveness of three different methods in decreasing pain during venipuncture in children: ball squeezing, balloon inflating and distraction cards. J Clin Nurs. 2016 Aug;25(15-16):2328-35. doi: 10.1111/jocn.13321. Epub 2016 Apr 26. PMID 27112434